CLINICAL TRIAL: NCT07263880
Title: Efficacy and Safety of Therapeutic Application of Clostridium Butyricum in Patiens With Stenosing Crohn's Disease: a Pilot Study
Brief Title: Clostridium Butyricum in Stenosing Crohn's Desease
Acronym: AUTOCD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: San Giovanni Addolorata Hospital (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Cristiano Pagnini, MD, PhD, San Giovanni Addolorata Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AUTOCD01
Record Dates: First submitted 2025-09-27; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease (CD)
Keywords: Clostridium butyricum, autophagy
MeSH Terms: conditions — Crohn Disease | interventions — Trehalose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C. butyricum (Experimental): Clostridium butyricum CBM 588 (27 x 10^5 CFU/day)
  Interventions: Dietary Supplement: Clostridum Butyricum Capsule
- Trehalose (Active Comparator): Threhalose (30g/day)
  Interventions: Dietary Supplement: Trehalose
- C butyricum + trehalose (Experimental): C. butyricum (27 x 10^5 CFU/day) + trehalose (30 g/day)
  Interventions: Dietary Supplement: Clostridum Butyricum Capsule; Dietary Supplement: Trehalose
- placebo (No Intervention): Patients with no treatment

INTERVENTIONS:
Dietary Supplement: Clostridum Butyricum Capsule — Administration of C. butyricum tablets (3 + 3 per day, 27 x 10^5 CFY/day)
  Arms: C butyricum + trehalose; C. butyricum
Dietary Supplement: Trehalose — Administration of trehalose at 30 g per day
  Arms: C butyricum + trehalose; Trehalose

SUMMARY:
Crohn's disease is a condition of unknown etiology with an immune-mediated pathogenesis. The subgroup of Crohn's disease with a stricturing phenotype represents a particular challenge for clinicians, as currently no effective medical therapies are available for the prevention or treatment of fibrosis. Autophagy is a key mechanism in the regulation of cellular homeostasis, and preliminary reports from our group and others have suggested a potential role in the pathogenesis of fibrostenotic complications in Crohn's disease.

The next-generation probiotic Clostridium butyricum has recently been proposed as a treatment option in several conditions, including inflammatory bowel diseases (IBD). Its beneficial effects are mainly exerted through the production of butyric acid, which in turn plays important roles at the intestinal mucosal level, including the stimulation of autophagy. The possibility of stimulating autophagy in patients with stricturing Crohn's disease may represent a promising therapeutic approach for the prevention and treatment of fibrosis.

This study involves the collection of biopsy and blood samples from 40 patients with stricturing Crohn's disease undergoing colonoscopy. In the two months preceding colonoscopy, patients will be randomized into four groups:

Patients treated with C. butyricum

Patients treated with the autophagy stimulator trehalose

Patients treated with C. butyricum + trehalose

Patients treated with placebo

Laboratory analyses will be performed on biopsy and blood samples to evaluate and quantify molecular mediators involved in inflammation, fibrosis, and autophagy.

DETAILED DESCRIPTION:
Crohn's disease is a chronic, relapsing inflammatory bowel disease with unknown etiology, involving immune dysregulation and microbiota alterations. Stricturing disease (Montreal B2 phenotype) represents a major unmet therapeutic need, as no pharmacological therapies are currently available for intestinal fibrosis, which is often managed surgically.

Autophagy, a key regulator of cellular homeostasis, has been linked to Crohn's disease pathogenesis, with genetic studies identifying polymorphisms in autophagy-related genes. Impaired autophagy may exacerbate inflammation, oxidative stress, and tissue damage. Preliminary data from our group show reduced autophagy in patients with stricturing Crohn's disease compared to those with inflammatory phenotype or healthy controls.

Clostridium butyricum, a next-generation probiotic with strong butyrate-producing activity, exerts anti-inflammatory and mucosal protective effects partly through stimulation of autophagy. Its use may represent a novel therapeutic approach to prevent or mitigate fibrostenotic complications in Crohn's disease.

This is a non-profit, interventional clinical pilot study enrolling 40 patients with stricturing Crohn's disease (B2, Montreal classification; localization L2 or L3). Patients undergoing clinically indicated colonoscopy will be randomized to one of four groups to receive for two months prior to the procedure:

1. C. butyricum supplementation
2. Trehalose supplementation (a known autophagy inducer)
3. Combined C. butyricum + trehalose
4. Placebo During colonoscopy, routine biopsies will be obtained, with two additional samples collected for research purposes, along with peripheral blood samples. Laboratory analyses will focus on molecular mediators of inflammation, fibrosis, oxidative stress, and autophagy pathways.

The primary objective is to test the hypothesis that C. butyricum is safe and capable of stimulating local autophagic processes in the intestinal mucosa of patients with stricturing Crohn's disease.

Secondary objectives include evaluating autophagy-related pathways (inflammation, fibrosis, ROS production, NADPH oxidase activity) and comparing outcomes across the four treatment groups. Laboratory procedures will be used to evaluate and quantify, in bioptic and blood samples autophagy, inflammation, fibrosis, and oxidative stress.In particular, autophagy will be evaluated by measurement of the mucosal autophagic markers LC3b-II and p62. Inflammation will be evaluated by measuring the expression of pro-inflammatory cytokines (TNFα, IFNγ, IL-17, and COX2), quantifying mRNA by real-time (RT)- PCR with specific primers. Fibrosis will be evaluated by quantification of mRNA of the related genes Col1a1, α-sma, Snail1, Snail2, TGFβ. Finally, oxydative stress levels will be evaluated by measuring serum markers such as sNOX2-dp, H2O2, and serum hydrogen peroxide (H2O2) breakdown activity (HBA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a confirmed diagnosis of Crohn's disease (established according to clinical, endoscopic, histological, and radiological criteria in line with current Italian and European guidelines), with a stricturing phenotype (B2 according to the Montreal classification), determined based on the patient's clinical history and instrumental examinations, with disease localized to the right colon or ileocecal region, followed at the Inflammatory Bowel Disease Outpatient Clinic of the Gastroenterology and Digestive Endoscopy Unit, in whom a colonoscopy with biopsies has been scheduled for clinical indication (disease reassessment, flare-up, or follow-up).
* Patients aged ≥18 and ≤85 years.
* Patients either not receiving any specific immunomodulatory therapy for Crohn's disease or undergoing treatment with mesalazine or sulfasalazine.
* Patients who have been adequately informed about the study protocol and who have understood and voluntarily signed the informed consent form.

Exclusion Criteria:

* Other acute or chronic inflammatory bowel diseases (e.g., diverticulitis, infectious colitis, ulcerative colitis).
* Patients receiving treatment for Crohn's disease with immunosuppressive drugs (thiopurines, methotrexate, cyclosporine), biologics (anti-TNFα, vedolizumab, ustekinumab), oral antiJAK or oral/intravenous corticosteroids.
* Immunological or rheumatologic diseases.
* Current or past malignancies.
* Active infections.
* History of organ transplantation.
* Current treatments with pharmacological agents known to significantly modulate the autophagic process.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of C. butyricum in stimulating autophagy | 2 months
  We evaluate the stimulation of autophagy measuring the mucosal expression and production of the molecular markers LC3 b II and p62 after treatment with C. butyricum
Safety of administration of C. butyricum | 2 months
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of C. butyricum in Crohn's disease patients will be evaluated by adverse event monitoring and reporting

SECONDARY OUTCOMES:
Treatment effect comparison | 2 months
  Comparation of the effect on autophagy induction (as mesured by LC3b-II and p62 mucosal production and expression), inflammatory (TNFα, IFNγ, IL-17 and COX2) and fibrosis (Col1a1, α-sma, Snail1, Snail2, TGFβ) markers in C. butyricum, trehalose, and C. butyricum+trehalose group
Oxydative stress measurement and comparation | 2 months
  Measurement and comparation of serum oxydative stress markers (sNOX2-dp, H2O2, and serum hydrogen peroxide [H2O2] breakdown activity - HBA) in the groups

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni Addolorata Hospital, Roma, Italy